CLINICAL TRIAL: NCT07135362
Title: The Efficacy Evaluation of Bifidobacterium Animalis Subsp. Lactis TCI604 Probiotic on Intestinal Function Improvement
Brief Title: The Efficacy Evaluation of TCI604 Probiotic on Intestinal Function Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202409097RSE
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Constipation; Intestinal Functional Disorder
Keywords: Bifidobacterium animalis subsp. lactis
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Taking 1 sachet of the testing sample with water every morning before breakfast for 4 consecutive weeks
  Interventions: Dietary Supplement: Placebo
- TCI604 probiotics (Experimental): Taking 1 sachet of the testing sample with water every morning before breakfast for 4 consecutive weeks
  Interventions: Dietary Supplement: TCI604 probiotics

INTERVENTIONS:
Dietary Supplement: TCI604 probiotics — TCI604 probiotics sachet
  Other Names: Bifidobacterium animalis subsp. lactis TCI604
  Arms: TCI604 probiotics
Dietary Supplement: Placebo — Placebo sachet
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate whether the TCI604 probiotics has the potential to enhance human gut function and alleviate constipation.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects aged 18 to 65 who are willing to sign the informed consent form;
* Diagnosed with functional constipation as assessed by a physician;
* Non-pregnant females who agree to use physical contraceptive methods during the study period (e.g., condoms, intrauterine devices);
* No history of organ transplantation, epilepsy or seizures, liver or kidney disease, malignancy, psychiatric disorders, alcohol or drug abuse, or other major organic diseases (as determined by medical history).

Exclusion Criteria:

* Use of probiotics, gastrointestinal health supplements, medications, or antibiotics within 30 days prior to the study;
* Presence of chronic gastrointestinal diseases (e.g., irritable bowel syndrome [IBS], inflammatory bowel disease [IBD], Crohn's disease, celiac disease, bowel control problems/fecal incontinence, pancreatitis, peptic ulcers, colorectal cancer, short bowel syndrome, ulcerative colitis);
* History of gastrointestinal or major surgery;
* Lactose intolerance;
* Chronic diarrhea;
* Pregnant or breastfeeding women;
* Known allergy to any components of the study product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The change of stool form | Week 0 (Baseline), Week 2, Week 4
  The stool type will be assessed by The Bristol Stool Form Scale (BSFS). The BSFS is a scale that classifies stools, ranging from the hardest (type 1) to the softest (type 7).
The change of bowel movement and gastrointestinal discomforts | Week 0 (Baseline), Week 2, Week 4
  The Gastrointestinal Symptom Rating Scale (GSRS) will be utilized to assess the bowel movement and gastrointestinal discomforts. The GSRS consists of 15 items, each rated on a 7-point Likert scale. A higher score indicates more severe and frequent symptoms.The total GSRS score is calculated by taking the average score of the five symptom categories- Reflux, Abdominal Pain, Indigestion, Diarrhea, and Constipation- summing them up, and then dividing the total by five to obtain the overall mean score.

SECONDARY OUTCOMES:
The change of intestinal microbiota | Week 0 (Baseline), Week 4
  Collect participant's feces for bacterial analysis. Intestinal microbiota will be assessed by Next Generation Sequencing (NGS).
The change of serum Interleukin-6 level | Week 0 (Baseline), Week 4
  A fasting blood sample will be collected for Interleukin-6 (IL-6) testing using an Enzyme-Linked Immunosorbent Assay kit.
The change of serum Interleukin-8 level | Week 0 (Baseline), Week 4
  A fasting blood sample will be collected for Interleukin-8 (IL-8) testing using an Enzyme-Linked Immunosorbent Assay kit.
The change of serum Interleukin-10 level | Week 0 (Baseline), Week 4
  A fasting blood sample will be collected for Interleukin-10 (IL-10) testing using an Enzyme-Linked Immunosorbent Assay kit.
The change of serum Interleukin-17A level | Week 0 (Baseline), Week 4
  A fasting blood sample will be collected for Interleukin-17A (IL-17A) testing using an Enzyme-Linked Immunosorbent Assay kit.
The change of blood High-sensitivity C-Reactive Protein level | Week 0 (Baseline), Week 4
  Venous blood samples will be collected to measure concentrations of High-sensitivity C-Reactive Protein.
The change of serum Lipopolysaccharide binding protein level | Week 0 (Baseline), Week 4
  A fasting blood sample will be collected for Lipopolysaccharide testing using an Enzyme-Linked Immunosorbent Assay kit.
The change of serum neopterin level | Week 0 (Baseline), Week 4
  A fasting blood sample will be collected for neopterin testing using an Enzyme-Linked Immunosorbent Assay kit.
The change of intestinal fecal loading | Week 0 (Baseline), Week 4
  Intestinal fecal loading will be evaluated using abdominal X-ray imaging.

OTHER OUTCOMES:
The change of Body weight | Week 0 (Baseline), Week 4
  Body weight will be assessed by Body Composition Analyzer. Unit: kg
The change of Body Mass Index | Week 0 (Baseline), Week 4
  Body Mass Index (BMI) level will be assessed by Body Composition Analyzer. Unit: kg/cm^2
The change of Percent Body Fat | Week 0 (Baseline), Week 4
  Percent Body Fat will be assessed by Bioelectrical Impedance Analysis (BIA) method. Unit: Percent
The change of Visceral Fat Level | Week 0 (Baseline), Week 4
  Visceral Fat Level will be assessed by Bioelectrical Impedance Analysis (BIA) method. Unit: arbitrary unit
The change of waist and hip circumference | Week 0 (Baseline), Week 4
  Waist and hip circumference will be assessed by measuring tape.
The change of blood pressure | Week 0 (Baseline), Week 4
  Systolic pressure and diastolic pressure will be assessed by sphygmomanometer.
The change of blood lipids profiles | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure concentrations of total cholesterol, High Density Lipoprotein Cholesterol, Low Density Lipoprotein Cholesterol, and triglyceride.
The change of blood liver function biomarkers (AST, ALT) | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure concentrations of liver function biomarkers.
The change of blood renal function biomarkers (creatinine, BUN) | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure concentrations of renal function biomarkers.
The change of blood fasting glucose level | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure concentrations of fasting glucose level.
The change of blood cells counts | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure the blood cells counts, including white blood cell (WBC) count/automated differential, red blood cell (RBC) count, platelet count. Unit: count/uL
The change of hemoglobin | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure the hemoglobin. Unit: g/dL
The change of hematocrit | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure the hematocrit. Unit: %
The change of mean corpuscular volume | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure the mean corpuscular volume (M.C.V). Unit: fl
The change of mean corpuscular hemoglobin concentration | Week 0 (Baseline), Week 4
  Venous blood will be sampled to measure the mean corpuscular hemoglobin concentration (M.C.H.C). Unit: g/dL

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Shiun Tsai, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan